CLINICAL TRIAL: NCT04848272
Title: Inhibition of Plasma Kallikrein as a New Therapy for Lung Injury
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: St Vincent's Institute of Medical Research (Other)
Responsible Party: Principal Investigator, Duncan Campbell, Associate Professor, St Vincent's Institute of Medical Research
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SVI-01
Record Dates: First submitted 2021-04-13; First posted 2021-04-19 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Lung Injury
MeSH Terms: conditions — Lung Injury | interventions — lanadelumab

STUDY DESIGN:
Intervention Model Description: Open-label placebo-controlled dose-escalation Phase 1 study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Saline control (Placebo Comparator): Saline control
  Interventions: Other: Saline control
- Lanadelumab 30 mg (Experimental): Lanadelumab 30 mg
  Interventions: Drug: Lanadelumab
- Lanadelumab 100 mg (Experimental): Lanadelumab 100 mg
  Interventions: Drug: Lanadelumab
- Lanadelumab 300 mg (Experimental): Lanadelumab 300 mg
  Interventions: Drug: Lanadelumab

INTERVENTIONS:
Drug: Lanadelumab — Monoclonal antibody that targets active plasma kallikrein
  Other Names: Takhzyro
  Arms: Lanadelumab 100 mg; Lanadelumab 30 mg; Lanadelumab 300 mg
Other: Saline control — Saline control
  Arms: Saline control

SUMMARY:
Phase 1 study investigating safety of lanadelumab administration to patients with lung injury

DETAILED DESCRIPTION:
This study will investigate the safety of inhibition of plasma kallikrein by lanadelumab administration in patients with lung injury.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years admitted to the ICU with primary diagnosis of lung injury. The criteria for the diagnosis of lung injury include five principal elements: hypoxemia (blood oxygen saturation (PaO2) ≤92% when breathing ambient air, ratio of PaO2 to the fraction of inspired oxygen (FiO2) ≤300), diffuse pulmonary infiltrates on chest radiographs, decreased lung compliance, and the absence of congestive heart failure.
* Both males and females will be recruited in the proportion in which they are admitted to the ICU with lung injury.
* Arterial cannula in place as part of usual care for the measurement of blood gases.
* Patients may or may not be intubated and mechanically ventilated.
* Able to provide informed consent, or if unable to do so, a responsible person:

medical treatment decision maker is available (by telephone if necessary) who can be approached to seek consent.

Exclusion Criteria:

* Other causes of lung infiltrates: pulmonary oedema, alveolar haemorrhage, adverse drug reactions, radiation injury and the idiopathic pneumonitis syndrome.
* Significant dysfunction of non-pulmonary organs in the opinion of the treating ICU consultant.
* Death is deemed imminent or inevitable or there is underlying disease with a life expectancy of less than 90 days.
* Previously enrolled in this study.
* Enrolled in another study.
* Usually receives home oxygen.
* Usually receives any type of assisted ventilation at home. e.g. continuous positive airway pressure for obstructive sleep apnoea.
* Pregnant or might be pregnant. Women aged 18 to 49 are excluded unless there is documented menopause, hysterectomy or surgical sterilisation, or a pregnancy test is negative.
* Objection from the treating clinician.
* Consent refused by the patient or substitute decision maker.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-08-09 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events | 28 days
  Blood gases, pH, bicarbonate, carbon dioxide and lactic acid levels. If the participant is receiving mechanical ventilation, the ventilator settings will be constantly monitored.
  Chest X-ray, as indicated. Constant monitoring of haemodynamics (pulse rate, blood pressure) via an arterial cannula, use of vasoactive medications, and constant monitoring of ECG. Fluid balance, including urine output. Serum creatinine, electrolytes, liver function, creatinine kinase, FBE and coagulation will be measured daily or less frequently as decided by the treating team.
  If there is suspicion of infection, then appropriate samples will be taken for microbiological examination.
  Neurological function will be assessed several times per day.

SECONDARY OUTCOMES:
Blood bradykinin concentration | 0, 6, 12, and 24 hours
  Blood bradykinin concentration

CONTACTS AND LOCATIONS:
Locations (1):
- St Vincent's Hospital Melbourne, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
Anonymised individual participant data (IPD) available to other researchers
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After completion of study
Access Criteria: To be determined